CLINICAL TRIAL: NCT06881888
Title: Intranasal Delivery of Octreotide for Treatment of Diabetic Macular Edema
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Maria Grant, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-300011278
Record Dates: First submitted 2025-03-05; First posted 2025-03-18 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; Intranasal Octreotide; Octreotide; Diabetic Retinopathy
MeSH Terms: conditions — Diabetic Retinopathy | interventions — Octreotide; Pharmaceutical Preparations; DDMS

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Octreotide Arm (Active Comparator): Participants will receive the investigational drug, DDM-Octreotide, and administering intranasally in one nostril three times a day.
  Interventions: Drug: Octreotide (drug)
- Control Group (Placebo Comparator): The control group will receive a placebo nasal spray without the active ingredient, DDM-octreotide, and administering intranasally in one nostril three times a day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Octreotide (drug) — Participants will administer the DDM-octreotide nasal spray without priming in one nostril three times a day.
  Other Names: Octreotide and 1-O-n-Dodecyl-b-D-Maltoyranoside (DDM) (Intravail®)
  Arms: Octreotide Arm
Drug: Placebo — Participants will administer the placebo nasal spray without priming in one nostril three times a day.
  Arms: Control Group

SUMMARY:
Treatment of diabetic retinopathy (DR) and diabetic macula edema has included panretinal photocoagulation and intra ocular injections of anti-vascular endothelial growth factors (anti-VEGF) agents and steroids. Anti-VEGF therapy is currently the first-line treatment for proliferative diabetic retinopathies; however, this approach is ineffective in more than 30% of patients with diabetic retinal complications. Available evidence shows that subcutaneous (under the skin) injection of octreotide, a somatostatin analog, has potential therapeutic benefits in proliferative diabetic retinopathy (PDR) and diabetic macula edema (DME). This study thus seeks to determine the efficacy and safety of intranasal DDM-octreotide in the treatment of diabetic macula edema in individuals that are considered to be refractory to the current therapeutic options.

ELIGIBILITY:
Inclusion Criteria:

1. Age range 18-90
2. Clinical diagnosis of diabetic retinopathy with diabetic macular edema (defined as CST greater than 250 and presence of microglia/macrophages on OCT) with a visual acuity between 20/32 and 20/200.
3. Written informed consent is provided.
4. Males and females
5. Routine laboratory study results with bilirubin, aspartate aminotransferase and/or alanine aminotransferase, and creatinine within normal limits.

Exclusion Criteria:

1. History of difficult to control diabetes or hypertension
2. Eyes receiving laser photocoagulation in the last 6 months or intravitreous treatment for diabetic macular edema in the past 3 months.
3. Eye having undergone YAG capsulotomy in the last 3 months.
4. Having other ocular surgeries in the last 6 months (examples include but not limited to cataract surgery, scleral buckle, trabeculectomies, etc.).
5. All women of childbearing potential must have a negative urine pregnancy test at the Screening Visit and throughout the study. Sexually active women participating in the study must use a medically acceptable form of contraception.
6. Chronic infectious disease (e.g. HIV, HCV)
7. Positive urine β-hCG test day of visit or a serum beta-HCG test within 48 hours prior to the administration of intranasal octreotide.
8. Other ocular diseases or fundus diseases
9. Patients with a history of intolerance or hypersensitivity to octreotide or use of octreotide in the preceding 2 months.
10. Currently taking an anti-inflammatory medication (e.g. anti-inflammatory agents, glucocorticoids or other immune modulating medications);
11. Use of cyclooxygenase-2 (COX-2) inhibitors for < 6 months prior to study entry or dose changes after study entry. Limited as-needed use is permitted prior to study entry but not during the study.
12. Use of statins that cross the blood brain barrier such as atorvastatin will not be permitted during the study as they have been shown to reduce levels of pro-inflammatory cytokines.
13. Any degree of hepatic or renal insufficiency that in the Investigator's judgement would pose a safety risk for treatment with octreotide.
14. Patients who based on history or mental status examination have a significant risk of committing suicide, or who are homicidal or violent and who are in the Investigator's opinion in significant imminent risk of hurting others.
15. Patients who have a medical condition that, in the Investigator's opinion, would expose them to an increased risk of a significant adverse event or interfere with assessments of safety and efficacy during the course of the trial.
16. Patients with a current known infection or who are acutely ill.
17. Patients with an autoimmune disease (i.e., Lupus, Rheumatoid Arthritis).
18. Patients with thyroid disorders unless euthyroid at screening.
19. Patients with cancer not in remission.
20. Inability to tolerate or intranasal administration of investigated drug and experiences severe irritation or sneezing.
21. Inability to attend scheduled study visits, plans for family relocation during the study, or any other criteria that the investigator may determine to be associated with inability to complete the study.
22. Limited mental capacity rendering the subject unable to provide written informed consent or comply with evaluation procedures.
23. History of recent alcohol or drug abuse or noncompliance with treatment or other experimental protocols.
24. Use of any investigational drug within 30 days prior to the baseline visit.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-08-31 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in macular central subfield thickness | Up to one month.
  Participants will have an optical coherence tomography at each visit that will measure macular central subfield thickness. Measuring the change at their baseline appointment and each additional study visit.
Change in best corrected visual acuity | Up to one month.
  Each participant will have best corrected visual acuity measured by Early Treatment of Diabetic Retinopathy study (ETDRS) chart. Enter the full scale.
Change in microglia on retinal surface | Up to one month
  Each participant will have an optical coherence tomography angiography scan measuring the quantity of microglia on the retinal surface.
Changes in retinal peripheral capillary free zone | up to one month
  Each participant will have optical coherence tomography angiography and measure differences in retinal peripheral capillary free zone.
Changes in retinal foveal avascular zone | up to one month
  Each participant will have optical coherence tomography angiography and measure differences in retinal foveal avascular zone.
Changes in retinal capillary density | up to one month
  Each participant will have optical coherence tomography angiography and measure differences in retinal capillary density.
Changes in retinal non-perfusion zones | up to one month
  Each participant will have optical coherence tomography angiography and measure differences in retinal non-perfusion zones.

SECONDARY OUTCOMES:
Changes in serum insulin like growth factor -1 (IGF-1) levels | up to one month.
  Each participant will have serum IGF-1 levels measured.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Grant, MD, FARVO, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Undecided